CLINICAL TRIAL: NCT03179306
Title: Cervix Image Sharing Protocol (CISP)
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999917098; 17-C-N098
Record Dates: First submitted 2017-06-06; First posted 2017-06-07 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Cervical Cancer; Cervical Abnormalities
Keywords: Cervix; HPV; Imaging; Costa Rica
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Samples: de-identified images and clinical data from NCI studies.

SUMMARY:
The Clinical Epidemiology Unit in the Clinical Genetics Branch of the Division of Cancer Epidemiology, NCI has a strong interest in fostering cervical cancer prevention solutions for all kinds of settings, including lowresource ones that rely on development of robust, low-cost screening and triage tools. Therefore, to support development of algorithms for cervical image recognition software, NCI seeks to share digital cervical images and accompanying clinical data from our large epidemiological studies on HPV and cervical cancer screening with interested and qualified image analysis researchers. To accommodate the many researchers that are interested, we have created this standard protocol to describe a unified process for sharing deidentified cervical images and accompanying de-identified clinical data from the following NCI studies: Costa Rican Natural History Study of HPV and Cervical Neoplasia , ASCUS LSIL Triage Study-- ALTS , SUCCEED and Costa Rica Vaccine Trial .

DETAILED DESCRIPTION:
The Clinical Epidemiology Unit in the Clinical Genetics Branch of the Division of Cancer Epidemiology, NCI has a strong interest in fostering cervical cancer prevention solutions for all kinds of settings, including lowresource ones that rely on development of robust, low-cost screening and triage tools. Therefore, to support development of algorithms for cervical image recognition software, NCI seeks to share digital cervical images and accompanying clinical data from our large epidemiological studies on HPV and cervical cancer

screening with interested and qualified image analysis researchers. To accommodate the many researchers that are interested, we have created this standard protocol to describe a unified process for sharing deidentified cervical images and accompanying de-identified clinical data from the following NCI studies: Costa Rican Natural History Study of HPV and Cervical Neoplasia , ASCUS LSIL Triage Study-- ALTS , SUCCEED and Costa Rica Vaccine Trial .

ELIGIBILITY:
* This protocol will include de-identified images and clinical data from NCI studies.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: collection of images and data from other NCI studies
Sampling Method: Non-Probability Sample
Enrollment: 27084 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-04-22 (Actual)

PRIMARY OUTCOMES:
Cervical intraepithelial neoplasia grade 3 (CIN3) or worse. | Occurrence at enrollment or during follow-up.
  The identification of CIN3 or cancer in histopathology analyses of biopsy and cervical excisional specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Julia C Gage, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States